CLINICAL TRIAL: NCT05077657
Title: Safe Surveillance of PCI Under Mechanical Circulatory Support With the Saranas Early Bird Bleed Monitoring System
Acronym: SAFE-MCS
Status: Completed | Type: Observational
Sponsor: Saranas, Inc. (Industry)
Collaborators: Proxima CRO (Industry); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Other Study IDs: PVP012
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single-Arm: This is a multi-center, single arm, open-label study to evaluate the safety of complex high-risk PCI using Impella and surveillance with the Saranas Early Bird Bleed Monitoring System (EBBMS).
  Interventions: Device: Early Bird® Bleed Monitoring System; Device: Impella®

INTERVENTIONS:
Device: Early Bird® Bleed Monitoring System — The Early Bird Bleed Monitoring System is used in endovascular procedures to monitor and detect internal bleeding complications in real-time.
Device: Impella® — Impella is an FDA-approved percutaneous heart pump indicated for patients with severe coronary artery disease requiring high-risk PCI.

SUMMARY:
The objective of this study is to establish the safety of complex high-risk Percutaneous Coronary Intervention (PCI) using Mechanical Circulatory Support (MCS) and surveillance with the Saranas Early Bird Bleed Monitoring System (EBBMS).

DETAILED DESCRIPTION:
To demonstrate that patients undergoing complex high-risk PCI using MCS and surveillance with the Saranas Early Bird Bleed Monitoring System will have relative incidence rate reduction of access site related BARC type III or V bleeding. An optimal outcome will show a a reduction in access-site related bleeding rate when using MCS with the Saranas EBBMS in high-risk PCI patients compared to historical incidence rate.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Planned complex high-risk PCI using MCS with Impella from a femoral access and use of Saranas Early Bird Bleed Monitoring System
* The study patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent as approved by the institutional review board of the respective clinical site.

Exclusion Criteria:

* Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
* Active bleeding
* Incapacity to access safely femoral artery or femoral vein
* Significant femoral, iliac, abdominal, or thoracic aortic disease which precludes placement of MCS
* Anemia (Hgb <9 g/dL), thrombocytopenia (Plt <50,000 cell/mL), history of bleeding diathesis or coagulopathy, or hypercoagulable states
* Active infection not controlled with antibiotic therapy
* Currently pregnant or women of child-bearing potential without documented negative pregnancy test
* Estimated life expectancy < 24 hours
* Patient is in cardiogenic shock at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing complex high-risk percutaneous coronary intervention (PCI) with mechanical circulatory support (MCS) via Impella® and transfemoral arterial approach will be enrolled. The Saranas Early Bird Bleed Monitoring System will be used in the ipsilateral femoral vein to monitor bleeding events after MCS removal.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Incidence of access site related BARC type III or V bleeding | Within 24 hours

SECONDARY OUTCOMES:
Incidence of activation of each Saranas Early Bird level 1, 2 and 3 indicator | Within 24 hours
Incidence of all BARC type III or V bleeding | Within 24 hours

OTHER OUTCOMES:
Access site related bleeding complications | Within 24 hours
  Safety Endpoint
Access site related vascular complications | Within 24 hours
  Safety Endpoint
Access site related blood transfusions | Within 24 hours
  Safety Endpoint
Non-access site related bleeding complications | Within 24 hours
  Safety Endpoint
Non-access site related vascular complications | Within 24 hours
  Safety Endpoint
Non-access site related blood transfusions | Within 24 hours
  Safety Endpoint
All blood transfusions | Within 24 hours
  Safety Endpoint
Hemoglobin drop | Within 24 hours
  Safety Endpoint
Death | Within 24 hours
  Safety Endpoint
Device and procedure-related adverse events | Within 24 hours
  Safety Endpoint
Serious adverse events | Within 24 hours
  Safety Endpoint
Serious adverse device effects | Within 24 hours
  Safety Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Mir Basir, DO, Principal Investigator — Henry Ford Hospital; Philippe Généreux, MD, Principal Investigator — Gagnon Cardiovascular Institute - Morristown Medical Center
Locations (11):
- United States (11):
  - St. Joseph Hospital / Arizona Heart, Phoenix, Arizona
  - Tucson Medical Center / PIMA Heart, Tucson, Arizona
  - Methodist Hospitals, Gary, Indiana
  - Ascension - St. John, Dearborn, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hackensack Meridian Health, Edison, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Northwell / Lenox Hill & Staten Island, New Hyde Park, New York
  - Memorial Hermann / UTH, Houston, Texas
  - St. Luke's / Texas Heart, Houston, Texas
  - Memorial Hermann NE / TCR Institute, Kingwood, Texas

IPD SHARING:
Plan to Share IPD: Undecided